CLINICAL TRIAL: NCT06045923
Title: Virologic and Immunologic Characteristics of Severe Mpox in Persons With Advanced HIV
Acronym: VIRISMAP
Status: Recruiting | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 7445
Record Dates: First submitted 2023-09-01; First posted 2023-09-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Monkeypox; HIV Infections; AIDS
MeSH Terms: conditions — Mpox, Monkeypox; HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Outpatient: 15 outpatients will be recruited from a single pre-determined clinical site (Columbia University)
- Inpatient: Up to 85 hospitalized patients will be recruited from other participating clinical sites

SUMMARY:
The purpose of this study is to examine the extent of mpox viral spread and immunologic markers in people with advanced HIV. Study findings will enhance knowledge of mpox pathogenesis in severely immunocompromised people, which can inform treatment and prevention of severe illness and deaths associated with mpox in people with advanced HIV.

DETAILED DESCRIPTION:
Primary objective:

Describe the relationship between the systemic immunologic response and the persistence and replication competence of mpox virus at rash lesions, in blood, and at mucosal sites over the course of mpox illness among patients with advanced HIV.

Secondary objectives:

* Describe the association between clinical outcomes and virologic and immunologic parameters among patients with severe mpox and advanced HIV.
* Survey for emergence of antiviral drug resistance among MPXV isolates collected over time during mpox illness among patients with advanced HIV.
* Characterize the effects of antivirals to treat mpox and/or HIV infection on virologic and immunologic parameters among patients with mpox and advanced HIV.
* Assess persistence and replication competence of mpox virus in the oropharynx and rectum over the course of mpox illness among patients with advanced HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years; AND
* HIV infection with CD4 count < 200 cells/uL; AND
* Probable or confirmed mpox (does NOT need to be a new diagnosis); AND
* Hospitalized while symptomatic from mpox, for reasons other than (or in addition to) infection prevention and control

Exclusion Criteria:

* Inability of the individual or appropriate proxy to provide informed consent.
* In the judgment of the clinical treating team, has a medical condition or other factor that might affect their ability to participate in the evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are hospitalized in the United States with probable/confirmed mpox and HIV with CD4 count < 200 cells/uL.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Monkeypox viral persistence | While hospitalized, for up to 12 months
  Monkeypox virus persistence in different sample types (including lesion, oropharyngeal, and rectal swabs; blood) over the course of illness
Monkeypox viral viability | While hospitalized, for up to 12 months
  Monkeypox virus viability in different sample types (including lesion, oropharyngeal, and rectal swabs; blood) over the course of illness
Immune response | While hospitalized, for up to 12 months
  Cytokine and chemokine profile over the course of illness

SECONDARY OUTCOMES:
Clinical outcome | Up to 12 months
  Duration of illness from mpox
Clinical outcome | Up to 12 months
  Duration of hospitalization with mpox
Clinical outcome | Up to 12 months
  Duration of critical illness due to mpox
Clinical outcome | Up to 12 months
  Mpox lesion burden
Clinical outcome | Up to 12 months
  Mortality
Clinical outcome | Up to 12 months
  Characterization of co-infections
Monkeypox virus resistance | While hospitalized, for up to 12 months
  Assess Monkeypox virus isolates for resistance to available therapeutics over the course of illness

CONTACTS AND LOCATIONS:
Overall Officials: Agam Rao, MD, Principal Investigator — Centers for Disease Control and Prevention; Irini Sereti, MD, Study Director — National Institutes of Health (NIH); Faisal Minhaj, Pharm.D., Study Director — Centers for Disease Control and Prevention; Shama Cash-Goldwasser, MD, Study Director — Centers for Disease Control and Prevention; Jesse OShea, MD, Study Director — Centers for Disease Control and Prevention; Christine Hughes, PhD, Study Director — Centers for Disease Control and Prevention; Brian Epling, MD, Study Director — National Institutes of Health (NIH); Katy Saliba, PhD, Study Director — National Institutes of Health (NIH); Jason Zucker, MD, Study Director — Columbia University; Sarah Reagan Steiner, MD, Study Director — Centers for Disease Control and Prevention; Sarah Park, MD, Study Director — Karius Laboratories
Locations (1):
- Centers for Disease Control and Prevention, Atlanta, Georgia, United States

REFERENCES:
- See also: VIRISMAP PowerPoint Presentation — https://www.cdc.gov/mpox/media/pdfs/2024/08/virismap-presentation.pdf